CLINICAL TRIAL: NCT06666309
Title: Optimizing PrEP Care Delivery Through Adaptive Intervention Strategies for Underserved Rural People Who Inject Drugs
Brief Title: Adaptive Intervention Strategies for HIV PrEP Care in Rural People Who Inject Drugs
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hilary L Surratt, PhD (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Hilary L Surratt, PhD, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 98939; R01DA061996-01 (NIH)
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-04

CONDITIONS: HIV Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Strengths Based Case Management - PrEP + Text Messaging (Experimental): Two session Strengths-based Case Management intervention delivered by a peer support specialist to individual clients in the syringe service program
  Interventions: Behavioral: SBCM-PrEP + Text Messaging
- CDC-PrEP + Text Messaging (Active Comparator): 1 session PrEP education following CDC guidelines delivered to individual clients in the syringe service program
  Interventions: Behavioral: CDC-PrEP + Text Messaging
- Strengths Based Case Management - PrEP + Text Messaging + Peer Transitional SBCM (T-SBCM) (Experimental): SBCM-PrEP + Text Messaging no response by end of month 1, and randomized to rup to 2 sessions of post-linkage transitional SBCM delivered by a peer support specialist
  Interventions: Behavioral: SBCM-PrEP + Text Messaging; Behavioral: T-SBCM
- Strengths Based Case Management - PrEP + Text Messaging + Mobile outreach (Experimental): SBCM-PrEP + Text Messaging no response by end of month 1, and randomized to up to 2 sessions of post-linkage field session visits delivered by a peer support specialist
  Interventions: Behavioral: SBCM-PrEP + Text Messaging; Behavioral: Mobile Outreach
- CDC-PrEP + Text Messaging + Peer Transitional SBCM (T-SBCM) (Other): CDC-PrEP + Text Messaging; no response by end of month 1, and randomized to rup to 2 sessions of post-linkage transitional SBCM delivered by a peer support specialist
  Interventions: Behavioral: CDC-PrEP + Text Messaging; Behavioral: T-SBCM
- CDC-PrEP + Text Messaging + Mobile outreach (Other): CDC-PrEP + Text Messaging no response by end of month 1, and randomized to up to 2 sessions of post-linkage field session visits delivered by a peer support specialist
  Interventions: Behavioral: CDC-PrEP + Text Messaging; Behavioral: Mobile Outreach

INTERVENTIONS:
Behavioral: SBCM-PrEP + Text Messaging — Two sessions Strengths-Based Case Management intervention adapted for HIV PrEP related educational content delivered to individual clients in the syringe service program setting
  Arms: Strengths Based Case Management - PrEP + Text Messaging; Strengths Based Case Management - PrEP + Text Messaging + Mobile outreach; Strengths Based Case Management - PrEP + Text Messaging + Peer Transitional SBCM (T-SBCM)
Behavioral: CDC-PrEP + Text Messaging — 1 session PrEP education based on CDC guidelines delivered to individual clients in syringe service program settings
  Arms: CDC-PrEP + Text Messaging; CDC-PrEP + Text Messaging + Mobile outreach; CDC-PrEP + Text Messaging + Peer Transitional SBCM (T-SBCM)
Behavioral: T-SBCM — Up to two post-linkage sessions of SBCM delivered by a peer support specialist in a format of the participants' choice (onsite, virtual/phone) in study month 2
  Arms: CDC-PrEP + Text Messaging + Peer Transitional SBCM (T-SBCM); Strengths Based Case Management - PrEP + Text Messaging + Peer Transitional SBCM (T-SBCM)
Behavioral: Mobile Outreach — Up to two in-person field session visits will be conducted by a peer support specialist for the purpose of offering direct support to arrange joint activities for overcoming identified barriers (e.g., transportation) to PrEP care initiation in study month 2.
  Arms: CDC-PrEP + Text Messaging + Mobile outreach; Strengths Based Case Management - PrEP + Text Messaging + Mobile outreach

SUMMARY:
During this 5-year study, stepped-care adaptive interventions will be deployed in three rural syringe service programs in a Sequential Multiple Assignment Randomized Trial (SMART) design to test the optimal intervention pathways for HIV PrEP uptake, defined as PrEP initiation (measured by dispensed prescription for oral PrEP) and persistence in PrEP care (measured by refill verification and biomarker confirmation). The study will be accomplished through three Specific Aims. AIM 1: Compare the relative effectiveness of adaptive interventions (AIs) that begin with Peer-led SBCM-PrEP versus those that begin with CDC-PrEP education plus text messaging (TM) on patient-level PrEP care outcomes (initiation and persistence) at 1-, 3- and 6-months; AIM 2: Estimate and rank the effectiveness of four embedded AIs on PrEP care outcomes at 3- and 6-months: (1) CDC-PrEP education, continue TM for responders, add Mobile Outreach for non-responders (NR); (2) CDC-PrEP education, continue TM for responders, add Peer transitional SBCM for NR; (3) Peer-led SBCM-PrEP, continue TM for responders, add Mobile Outreach for NR; (4) Peer-led SBCM-PrEP, continue TM for responders, add Peer transitional SBCM for NR. AIM 3: Across interventions, examine the effects of age, baseline injection frequency, perceived HIV risk, PrEP interest, SSP utilization patterns, and other factors, in predicting PrEP care outcomes at 1-, 3- and 6-months to inform optimally-tailored intervention strategy recommendations.

DETAILED DESCRIPTION:
Kentucky's HIV epidemic displays an especially profound and disproportionate impact among people who inject drugs (PWID): 14.8% of males and 54.2% of females newly diagnosed with HIV in 2021 have an injection drug use-related transmission factor, far exceeding the national average for this exposure category. A central pillar of Ending the HIV Epidemic (EHE) is the prevention of new HIV infections through scale up of Pre-Exposure Prophylaxis (PrEP) in key populations, including PWID. For PWID, PrEP uptake remains severely limited, and no evidence-based PrEP interventions specifically targeted for PWID are available. In the previous pilot in KY's Appalachian region, two brief, low-intensity interventions to promote linkage to co-located PrEP care in rural syringe service programs (SSPs) were successfully implemented, including a newly adapted strengths-based case management (SBCM-PrEP) intervention designed to address multi-level barriers to PrEP initiation. The pilot trial has demonstrated proof of concept for integrated PrEP care within rurally-located SSPs and high acceptability among PWID with high uptake of initial clinical interventions. Nevertheless, just 51% returned for test results, and 28% progressed to PrEP prescription, indicating that augmented intervention support is required to optimize PrEP uptake. The stepped-care Adaptive Interventions (AIs) to be tested respond directly to identified challenges in the pilot trial and the need for augmented support among initial non-responders. AIs have shown remarkable promise in diverse behavioral and medical conditions, including areas such as chronic lower back pain, risky drinking and violent behavior, reducing alcohol use, preventing suicidal behavior, and HIV treatment retention

ELIGIBILITY:
Inclusion Criteria:

* self-report of at least one occasion of injection drug use in the past month
* use of the SSP in the past 30 days
* expressed willingness to participate in a multi-session intervention and follow-up
* having an indication for PrEP in the past 6 months based on CDC guidelines

Exclusion Criteria:

* being HIV positive
* current PrEP care
* self-reported severe renal impairment and/or chronic HBV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants initiating PrEP | 1 month post-baseline
  Documented PrEP initiation, measured by dispensed prescription
Number of participants initiating PrEP | 3 months post-baseline
  Documented PrEP initiation, measured by dispensed prescription
Number of participants initiating PrEP | 6 month post-baseline
  Documented PrEP initiation, measured by dispensed prescription

SECONDARY OUTCOMES:
Linkage to PrEP Care | 1 month post-baseline
  Number of participants completing initial clinical evaluation for PrEP, measured by provider report
Linkage to PrEP Care | 3 month post-baseline
  Number of participants completing initial clinical evaluation for PrEP, measured by provider report
Linkage to PrEP Care | 6 month post-baseline
  Number of participants completing initial clinical evaluation for PrEP, measured by provider report
PrEP Persistence | 3 months post-baseline
  Number of participants receiving dispensed PrEP refill, measured by provider report/pharmacy verification.
PrEP Persistence | 6 months post-baseline
  Number of participants receiving Dispensed PrEP refill, measured by provider report/pharmacy verification.
PrEP Adherence | 3 months post-baseline
  Number of participants with Presence of PrEP (TFV) in blood sample
PrEP Adherence | 6 months post-baseline
  Number of participants with Presence of PrEP (TFV) in blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Hillary L Surratt, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - University of Kentucky, Lexington, Kentucky
  - Clay County Health Department, Manchester, Kentucky

IPD SHARING:
Plan to Share IPD: Yes
All Aim 1 and 2 de-identified REDCap survey data and clinical data extracts from report forms will be preserved and shared. We will not share participant locator information. Datasets will be shared as CSV files.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study team will submit a de-identified and cleaned survey and clinical dataset within 12 months after the last participant's study visit, or at acceptance of the primary outcomes paper for publication, whichever is first.
Access Criteria: De-identified survey and clinical data will be shared with controlled access in for general research use.